CLINICAL TRIAL: NCT04873063
Title: Explorative Study of the Safety/Tolerability of Beclomethasone Dipropionate Suppositories: Evaluation of Systemic Bioavailability and Effects on 24-Hour Plasma Cortisol Profile of 6 mg Delivered Once Daily Versus 3 mg Delivered Twice Daily in Healthy Adult Male Volunteers
Brief Title: Evaluation of Systemic Bioavailability and Effects on 24-Hour Plasma Cortisol Profile of 6 mg Delivered Once Daily Versus 3 mg Delivered Twice Daily in Healthy Adult Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SOFAR S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: PSC DS BDP-Once 1
Record Dates: First submitted 2021-04-26; First posted 2021-05-05 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Healthy Adult Male Volunteers
MeSH Terms: interventions — Beclomethasone

STUDY DESIGN:
Intervention Model Description: Single-centre, randomized, double-blind, two-period, two-sequence, cross-over 7-day study.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference/Test (Experimental): * 3 mg BDP suppositories (R product) delivered twice daily for 7 days
  * Washout period (at least 7-day and preferably no more than 9 days)
  * 6 mg BDP suppositories (T product) delivered once daily in the morning for 7 days. Matching placebo suppository will be applied rectally once daily in the evening, on same days as the T product.
  Interventions: Drug: Beclomethasone dipropionate
- Test/Reference (Experimental): * 6 mg BDP suppositories (T product) delivered once daily in the morning for 7 days. Matching placebo suppository will be applied rectally once daily in the evening, on same days as the T product.
  * Washout period (at least 7-day and preferably no more than 9 days)
  * 3 mg BDP suppositories (R product) delivered twice daily for 7 days
  Interventions: Drug: Beclomethasone dipropionate

INTERVENTIONS:
Drug: Beclomethasone dipropionate — BDP 3 mg bid (R product) BDP 6 mg qd (T product)
  Other Names: Beclomethasone 17,21-dipropionate; BDP

SUMMARY:
Single-centre, randomized, double-blind, two-period, two-sequence, cross-over 7-day study.

This study is the first safety/tolerability evaluation of a product -suppository formulation containing 6 mg BDP (once daily dosing), a second-generation oral or rectal corticosteroids with high topical anti-inflammatory efficacy in the gut and minimal systemic bioavailability (BA).

BDP is marketed in different pharmaceutical formulations, including 3 mg suppositories, and approved for ulcerative proctosigmoiditis in the first attack or exacerbation phase at the dosage of 3 mg twice a day. For these reasons, a 6 mg suppository (Test - "T" product) is a scale-up of the 3 mg formulation (Reference - "R" product).

For locally-applied-locally acting drug products that result in quantifiable systemic availability due to absorption from the administration site, relative systemic BA is informative for safety, but also with respect to efficacy. Therefore, safety/tolerability of T is evaluated through a comparison to R.

DETAILED DESCRIPTION:
Primary objective is the evaluation of systemic safety of T, based on valid surrogate outcomes - systemic BA (relative BA) at the start of treatment (first 24 hours) and after 7 days of continuous treatment; effects on the hypothalamo-pituitary-adrenal axis (HPA) assessed based on 24-hour cortisol profile after 7 days of continuous treatment. This includes identification of subjects with cortisol levels <10 μg/dL at the last sampling point in the 24-hour cortisol profile (08:00 a.m. on Day 8). In such cases, identified subjects will undergo ACTH stimulation test in the morning of Day 9.

Secondary objective is the evaluation of safety/tolerability based on clinical and laboratory adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male, aged between 18 and 55 years. Healthy subjects are defined as individuals who are free from clinically significant illness or disease as determined by their medical history, physical examination, laboratory and other (e.g. ECG) tests.
* BMI 19.0 - 29.0 kg/m2;
* Signed and dated written informed consent of the subject to participate in the clinical study;
* The subject is willing to refrain from the use of illicit drugs and alcohol and to adhere to other protocol-stated restrictions while participating in the study;
* The subject is able to understand and comply with the protocol requirements and instructions and is likely to complete the study as planned;
* Non-smoker for at least 3 months.

Exclusion Criteria:

* Subject with a significant abnormality in the past and/or at the Screening that influences the present general health condition and requires pharmacological treatment during the study;
* History of serious allergic diseases, including allergy to medicinal products, which in opinion of the investigator, contraindicates participation to the trial;
* History of diseases of the alimentary tract, liver or kidneys that may influence absorption, distribution and elimination;
* History of average alcohol consumption;
* Hypersensitivity to BDP or study products inactive ingredients;
* Use of any pharmacological treatments (including high dose vitamins, lozenges, herbal and dietary supplements), with the exception of paracetamol ≤ 1 g/daily, within 15 days before the admission to the study Site in the Period 1;
* Use of steroids, anabolic or hormonal therapy within 3 months before the admission to the study Site in the Period 1;
* Laboratory indication of adrenocortical dysfunction;
* Blood loss exceeding 200 ml over the last 4 weeks before the day of Screening;
* Positive results to Sars Cov-2 nasopharyngeal swab;
* Positive results of HBsAg, anti-HCV, anti-HIV tests;
* Blood pressure: systolic >140mmHg or < 90mmHg, diastolic <60 mmHg or >90 mmHg during screening procedures;
* Subject who adhere to a special diet (e.g. low calories, vegetarian etc.);
* Consumption of products containing methylxanthines in the following average quantities: > 3 cups of 200 ml of strong coffee a day;
* Presence of metabolites of illicit drugs (opioids, cannabis) during screening procedures;
* Participation in other clinical trials during the 6 months preceding the study, counting from the day of last product administration.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax, morning; | Day 1 and Day 7 of each Period
  Peak exposure after the morning dose (Cmax, morning)
Pharmacokinetics - Cmax, evening; | Day 1 and Day 7 of each Period
  Peak exposure after the evening dose (Cmax, evening)
Pharmacokinetics - AUC0-24 | Day 1 and Day 7 of each Period
  • Total exposure over 24 hours (AUC0-24)
Pharmacokinetics - AUC0-12 | Day 1 and Day 7 of each Period
  • Total exposure during dosing interval - morning (AUC0-12)
Pharmacokinetics - AUC12-24 | Day 1 and Day 7 of each Period
  • Total exposure during dosing interval - evening (AUC12-24)
HPA-axis: 24-hour plasma cortisol - AUC0-24, cortisol | Baseline and Day 7 of each Period
  Area under the cortisol level-time curve over 24 hours (AUC0-24, cortisol). AUC will be determined for each subject/treatment at baseline and at Day 7 by the linear trapezoidal rule and ln-transformed.
  Ln(AUCs) will be used to determine intra-subject difference Day 7 - baseline that will be subject to analysis.
HPA-axis: 24-hour plasma cortisol - AUC0-12, cortisol | Baseline and Day 7 of each Period
  Area under the cortisol level-time curve over 12 hours after the morning dose (AUC0-12, cortisol).
  As above.
HPA-axis: 24-hour plasma cortisol - AUC12-24, cortisol | Baseline and Day 7 of each Period
  Area under the cortisol level-time curve over 12 hours after the evening dose (AUC12-24, cortisol).
  As above.
HPA-axis: 24-hour plasma cortisol - pAUC2-8, cortisol | Baseline and Day 7 of each Period
  Partial area under the cortisol level-time curve "covering" 3rd, 4th, 5th, 6th, 7th and 8th hour post morning dose (i.e., between 10:00 and 16:00 hours, that is, between sampling times at 2 and 8 hours post-dose) - a time period during which normal cortisol levels are still relatively high and the strongest suppression after morning dose could be expected (pAUC2-8, cortisol).
  As above.

SECONDARY OUTCOMES:
Pharmacokinetics - trough concentrations | Day 1 and Day 7 of each Period
  Trough concentrations for R (C12) and T (C24) dosing on Day 1 and Day 7 as well as morning pre-dose (C0)
Pharmacokinetics - Cmax morning/AUC0-12 ratio | Day 1 and Day 7 of each Period
  Ratio of the peak exposure after the morning dose to exposure over the subsequent 12 hours (illustrates absorption rate) (Cmax,morning/AUC0-12)
Pharmacokinetics - Tmax, morning | Day 1 and Day 7 of each Period
  Time to peak exposure after the morning dose (Tmax,morning)
Pharmacokinetics - Percent fluctuation (%PTF12) | Day 7 of each Period
  Day 7 - percent fluctuation over 12 hours after morning dose (%PTF12)
Pharmacokinetics - Percent fluctuation (%PTF24) | Day 7 of each Period
  Day 7 - percent fluctuation over 24 hours (%PTF24)
Pharmacokinetics - Accumulation ratio | Day 1 and Day 7 of each Period
  Accumulation ratio (Cmax,morning Day 7/Day 1; AUC0-24 Day 7/Day 1). Accumulation ratio will be estimated based on two outcomes: peak exposure after the morning dose (Cmax, morning) and total exposure over 24 hours (AUC0-24).
HPA axis - Number (proportion) of subjects with cortisol <10 μg/dL | Day 8 and 9 of each Period
  ACTH stimulation test results on the morning of Day 9 (first post-dosing day) dichotomized as "normal" or "abnormal"
HPA axis - Number/proportion of subjects with abnormal ACTH stimulation test. | Day 8 and 9 of each Period
  Number (proportion) of subjects with cortisol levels <10 μg/dL at 08:00 a.m. on Day 8 and number (proportion) of subjects with abnormal ACTH stimulation test results in the morning of Day 9 (should any subject be submitted).
HPA axis - 24-hour cortisol profile | Baseline and Day 7 of each Period
  24-hour cortisol profile: time-point-by-time-point differences Day 7 vs. baseline

OTHER OUTCOMES:
Safety - Adverse Events | From screening to follow up (approximately 59 days)
  Adverse events reporting
Safety - Laboratory values | At screening, before each period and at follow-up (+21 days after the end of Period 2)
  Incidence of abnormal laboratory test results (Urinalysis, biochemical and haematological tests performed)

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Ricerche Cliniche AOU Integrata di Verona - Policlinico Universitario G.B. Rossi, Verona, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR